CLINICAL TRIAL: NCT04389307
Title: Bladder Training With and Without Intravaginal Electrical Stimulation in Women With Idiopathic Overactive Bladder: A Prospective Randomised Controlled Trial
Brief Title: Intravaginal Electrical Stimulation in Idiopathic Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hakan Alkan, Clinical Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19892010-2019
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Idiopathic Overactive Bladder; Electrical Stimulation; Bladder Training
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Bladder Training - Control group (Other): Specific goals are to correct faulty habit patterns of frequent urination, improve control over bladder urgency, prolong voiding intervals, increase bladder capacity, reduce incontinence episodes and restore patient confidence in controlling bladder function
  Interventions: Other: Bladder Training
- Group 2: Bladder Training+Intra Vaginal Electrical Stimulation (Active Comparator): IVES was performed in lithotomy position via Enraf Nonius Myomed 632 device with a vaginal probe. IVES sessions were performed three times in a week, for 8 weeks. Every session lasted 20 minutes. The intervention comprised a 24-session treatment program of ES. The stimulation parameters were frequency at 10 Hz, a 5-10s work-rest cycle and 100 ms pulse width. The symmetric biphasic pulse wave could be delivered over a range of 0-100 mA. The intensity was controlled according to patients' discomfort level feedback
  Interventions: Other: Electrical stimulation (IVES); Other: Bladder Training

INTERVENTIONS:
Other: Electrical stimulation (IVES) — IVES sessions were performed three times in a week, for 8 weeks. Every session lasted 20 minutes. The intervention comprised a 24 session treatment program of IVES.
  Arms: Group 2: Bladder Training+Intra Vaginal Electrical Stimulation
Other: Bladder Training — Bladder Training

SUMMARY:
Overactive bladder (OAB) is a symptom complex defined as urgency, with or without urge urinary incontinence (UUI), usually with frequency and nocturia, in the absence of urinary tract infection. Currently, a wide range of therapeutic options exist for the treatment of OAB. These include first-line conservative (physical) therapies which focus on electrical stimulation (ES) and behavioral therapies such as lifestyle modifications, bladder training (BT), pelvic floor muscle training with or without biofeedback, second-line therapies which are pharmacologic, and third-line therapies which either neuromodulate or chemodenervate the bladder.

In clinical practice, BT and Intravaginal ES (IVES) are frequently used together in the treatment of women with OAB, but the evidences/results of the combined (BT+IVES) use of these two treatment options are so rare that they can be neglected in the literature. There is only one study including BT+ES treatment arm (one of the four treatment arms) in women with idiopathic OAB in the literature. In a study, BT+ES was not found to be effective both from BT alone and from the untreated control group. While interpreting the results of this study, it should be take into consideration that patients treated received relatively few treatment sessions (nine treatment sessions, once weekly) in this study. In addition, in the light of authors clinical experience, the investigators think that this issue is still open for research. Moreover, there is no recommendation on conservative combinations in the guidelines due to insufficient data.

This study is the first prospective randomized controlled trial that compares the efficacy of BT and BT plus IVES in women with idiopathic OAB. In this study, the investigators aimed to evaluate the efficacy of BT with and without IVES on incontinence-related QoL and clinical parameters in women with idiopathic OAB.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 with clinical diagnosis of idiopathic OAB
* Urodynamically diagnosed detrusor overactivity
* The strength of pelvic floor muscle 3/5 and more
* Able to give written, informed consent
* Able to understand the procedures, advantages and possible side effects
* Willing and able to complete the voiding diary and QoL questionnaire

Exclusion Criteria:

* History of conservative therapy (BT, ES) for OAB within 3 months
* Previously treated with antimuscarinics (within 4 weeks)
* Pregnancy or intention to become pregnant during the study
* Current vulvovaginitis or urinary tract infections or malignancy
* History of urogynecological surgery within 3 months
* Anatomic structural disorders of genital region that could not allow to apply the vaginal probe
* Having stage 2 or more according to the pelvic organ prolapse quantification
* Cardiac pacemaker or implanted defibrillator
* Neurogenic bladder, signs of neurologic abnormalities at objective examination; history of the peripheral or central neurologic pathology
* Ultrasonographic evidence of residual urine volume more than 100 ml
* Allergy to condom or lubricant gel that is used with perineometer/vaginal probe

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
incontinence episodes-incontinence related outcomes measures | 8 weeks
  Patients with a 50% or greater reduction in incontinence episodes were consider positive responders (number of voiding per day)

SECONDARY OUTCOMES:
frequency of voiding-incontinence related outcomes measures | 8 weeks
  it was used frequency from data with a bladder diary (number of voiding per day)
nocturia frequency- incontinence related outcomes measures | 8 weeks
  it was used nocturia from data with a bladder diary (number of voiding per night)
incontinence related quality of life questionnaire | 8 weeks
  (IIQ-7) (score)

CONTACTS AND LOCATIONS:
Locations (1):
- Hakan Alkan, Denizli, None Selected, Turkey (Türkiye)